CLINICAL TRIAL: NCT06906263
Title: Complications Related to the Anaesthesia During Airway Endoscopy in Children with Tracheostomy.
Status: Not yet recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ida Engqvist, Medical doctor, Principal Investigator, Karolinska Institutet
Other Study IDs: 2023-07493-01
Record Dates: First submitted 2025-03-18; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia Complication; Tracheostomy Complications; Children Receiving General Anesthesia
Keywords: Tracheostomy; Pediatric; Anesthesia complication; general anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children below 18yrs with tracheostomy undergoing follow-up with surveillance airway endoscopy: The children with tracheostomy undergoing follow-up with surveillance airway endoscopy under general anasthesia through the Long term intensive care unit (LIVA) at Karolinska Hospital Stockholm Sweden between jan 2025-dec 2026.

SUMMARY:
The goal of this observational study is to investigate the incidence of severe anaesthesiologic complications during anaesthesia in children with tracheostomy undergoing surveillance airway endoscopy. The main question it aims to answer is how common severe anaesteshiologic complications are in these patients and investigate if there is an association between severe anaesthesiologic complications and patient related factors.

Primary outcome: The incidence of severe anaesthesiologic complications in children with tracheostomy undergoing surveillance airway endoscopy.

Secondary outcome: The association between severe anaesthesiologic complications and patient related factors: age at tracheostomy, age at surveillance endoscopy, ventilator dependence, current and previously diagnosed tracheostomy related airway complications.

All children under 18 yrs. of age with a tracheostomy accepted for general anaesthesia undergoing surveillance airway endoscopy at the Long term Intensive Care unit at Karolinska University Hospital Stockholm Sweden will be eligable for inclusion. The anaesthesia will be conducted according to current practise and complications will recorded by the anaesthesiologist in charge. Participants may only be included once.

DETAILED DESCRIPTION:
Background:

Children with airway obstruction due to inborn malformations or trauma, or who have a chronic need for respiratory support due to lung- or neuromuscular diseases, may require a tracheostomy. A tracheostomy is a surgical opening of the trachea at the front of the neck to create an artificial airway, maintained with a tracheostomy tube. The Long-term Intensive Care Unit (LIVA) is a unit within Paediatric Perioperative Medicine and Intensive Care (BPMI) at Karolinska University Hospital. Since 1998, its primary task has been to care for children with tracheostomies from a large part of the country and it is the only unit of its kind in Scandinavia.

LIVA's follow-up of children with tracheostomies includes 1-2 surveillance airway endoscopies under anaesthesia per year. The endoscopies aim to early identify airway complications related to the tracheostomy tube. Complications, such as granulomas, infections, or bleeding, are often asymptomatic, and potentially lethal. There is no international nor national consensus regarding how often surveillance endoscopies should be performed. The possibility of individualizing the surveillance program based on risk factors has not been explored. Every anaesthesia carries a potential risk for the child. The incidence of complications related to the anaesthesia in children with tracheostomy undergoing airway endoscopy has not yet been investigated.

In this study the investigator aim at assessing the incidence of anaesthesia-related complications during the surveillance airway endoscopies. Understanding the anaesthesiologic risk associated with the endoscopies is important in weighing risk versus benefit with the current surveillance airway endoscopy program.

Main objective: To investigate the incidence of anaesthesiologic complications in children undergoing airway endoscopy as part of the surveillance program for children with tracheostomy.

Research outcomes:

Primary outcome: What is the incidence of severe anaesthesiologic complications in children with tracheostomy undergoing surveillance airway endoscopy? Secondary outcome: Is the risk for anaesthesia complications associated with patient related factors such as age, comorbidity and indication for tracheostomy?

Method: This is a prospective observational study. All children with tracheostomy undergoing follow-up through LIVA scheduled to undergo a surveillance endoscopy will be eligible for inclusion continued until 80 investigations have been performed or the 2 year investigation period has ended. Participants may only be included once. The anaesthesia is conducted according to current practice. Anaesthesia-related complications are recorded by the anaesthesiologist in charge through a standardized protocol including occurrences of hypoxemia, bronchospasm, aspiration, severe bradycardia and hypothermia, during anaesthesia and in the immediate postoperative period. Demographic data and information regarding risk factors with regards to anaesthesiologic complications are collected from patient charts. Ethical approval has been obtained, ref. no2023-07493-01.

ELIGIBILITY:
Inclusion Criteria:

All patients

1. under the age of 18yrs
2. with tracheostomy
3. undergoing surveillance airway endoscopy
4. approved for anesthesia

will be included once within the time frame of the study (2years).

Exclusion Criteria:

If other scheduled major surgery will take place in the same session or if the airway endoscopy is a non-elective emergency procedure, inclusion will not take place for that procedure. The same patient may however be eligible for inclusion at a later date, during the inclusion period, if subject to a subsequent airway endoscopy that meets the inclusion criteria.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children below 18yrs with tracheostomy undergoing follow-up with surveillance airway endoscopy in general anesthesia at the Long Term Intensive Care unit (LIVA) at Karolinska University Hospital in Stockholm Sweden will be studied. This includes a majority of the children with tracheostomy in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
severe anaesthesiologic complications | Perioperative
  The incidence of severe anaesthesiologic complications in children with tracheostomy undergoing surveillance airway endoscopy.

SECONDARY OUTCOMES:
Association between severe anaesthesiologic complications and patient related factors | Perioperative
  The association between severe anaesthesiologic complications and patient related factors: age at tracheostomy, age at surveillance endoscopy, ventilatory dependence, current and previously diagnosed tracheostomy related airway complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Perioperative Medicine and Intensive Care, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al Bahri K, Liu CC. Surveillance endoscopy in pediatric tracheostomy: A systematic review. Int J Pediatr Otorhinolaryngol. 2021 Jan;140:110533. doi: 10.1016/j.ijporl.2020.110533. Epub 2020 Dec 1. PMID 33296833
- [Background] Habre W, Disma N, Virag K, Becke K, Hansen TG, Johr M, Leva B, Morton NS, Vermeulen PM, Zielinska M, Boda K, Veyckemans F; APRICOT Group of the European Society of Anaesthesiology Clinical Trial Network. Incidence of severe critical events in paediatric anaesthesia (APRICOT): a prospective multicentre observational study in 261 hospitals in Europe. Lancet Respir Med. 2017 May;5(5):412-425. doi: 10.1016/S2213-2600(17)30116-9. Epub 2017 Mar 28. PMID 28363725
- [Background] Liu CC, Soares JJ, Elder L, Hill L, Abts M, Bonilla-Velez J, Dahl JP, Johnson KE, Ong T, Striegl AM, Whitlock K, Parikh SR. Surveillance endoscopy after tracheostomy placement in children: Findings and interventions. Laryngoscope. 2020 May;130(5):1327-1332. doi: 10.1002/lary.28247. Epub 2019 Oct 31. PMID 31670383